CLINICAL TRIAL: NCT01153776
Title: CT Coronary Angiography for the Detection of Reimplanted Coronary Lesions in Patients Who Had Undergone Arterial Switch Operation for Transposition of the Great Arteries
Brief Title: CT Coronary Angiography After Arterial Switch Operation
Acronym: SCANTGV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P070118; 2007-A00833-50 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: CT Coronary Angiography; Arterial Switch Operation
Keywords: Arterial switch operation; Transposition of the great arteries; Congenital heart diseases; CT coronary angiography
MeSH Terms: conditions — Transposition of Great Vessels; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 64-slice CT angiography (Experimental): 64-slice CT angiography
  Interventions: Procedure: 64-slice CT angiography

INTERVENTIONS:
Procedure: 64-slice CT angiography — the sensitivity and specificity of 64-slice CT angiography for the detection of lesions at the ostia and proximal segments of the reimplanted coronary arteries

SUMMARY:
The purpose of this study is to find a non-invasive alternative (with using ECG gated 64-slice CT angiography) to invasive coronary angiography for detecting coronary lesions in patients who had undergone arterial switch operation for transposition of the great arteries

DETAILED DESCRIPTION:
Objectives To find a non-invasive alternative (with using ECG-gated 64-slice CT angiography) to invasive coronary angiography for detecting coronary lesions in children who had undergone arterial switch operation for transposition of the great arteries.

Background Assessment of the integrity of reimplanted coronary arteries is crucial for long-term outcome after arterial switch operation for transposition of the great arteries. Non-invasive tests have limited accuracy for detecting coronary lesions, and invasive coronary angiography is usually required in this setting.

Materials and methods Patients (age 4 to 30 years old) who undergone arterial switch operation in neonate period are potentially eligible. They will be prospectively included in the study. They will have both examinations, their routine invasive coronary angiography and ECG-gated 64-slice CT angiography. The ability of CT to detect lesions of the ostia and proximal segments of the reimplanted coronary arteries was analyzed by blinded comparison to invasive coronary angiogram.

Expected results and clinical implications We expect to demonstrate that ECG-gated 64-slice CT angiography is safe and accurate for the detection of coronary lesions with a high sensitivity (expected sensitivity>95%) as compared to invasive angiography. In that condition, ECG-gated 64-slice CT angiography could replace the invasive coronary angiography for the follow-up of patients with reimplanted coronary arteries after arterial switch operation for transposition of the great arteries.

ELIGIBILITY:
Inclusion criteria :

* patients, age 4 to 30 years old, who had undergone arterial switch operation for transposition of the great arteries, are eligible.

Exclusion criteria :

* No consent
* Allergy to contrast agent (iodine contrast)
* Severe renal failure (clearance < 80ml/min/1.73m²)
* Severe arrhythmias
* Absence of medical care insurance
* Pregnancy
* Contre-indication to beta-blockers

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of 64-slice CT angiography for the detection of lesions at the ostia and proximal segments of the reimplanted coronary arteries | 30 MINUTES
  Sensitivity and specificity of 64-slice CT angiography for the detection of lesions at the ostia and proximal segments of the reimplanted coronary arteries
  Expected sensitivity > 95% Expected specificity > 95%

CONTACTS AND LOCATIONS:
Overall Officials: Ou Phalla, MCU Ph, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France